CLINICAL TRIAL: NCT02133859
Title: Feasibilty of Respiratory Monitoring With Adaptive Servoventilation (PaceWave™) to Predict Worsening of Heart Failure in Patients With Severe Heart Failure and Sleep-disordered Breathing
Brief Title: Adaptive Servo-ventilation Monitoring Study
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: MA220414
Record Dates: First submitted 2014-05-01; First posted 2014-05-08 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Heart Failure patients using ASV: Patients with chronic heart failure who are using or willing to use adaptive servo ventilation (ASV) therapy will be enrolled. Respiratory data will be collected from this group every 3 months over a 12 month period

SUMMARY:
Sleep disordered breathing is very common in patients with chronic heart failure with reported prevalence rates of 50-75%. Adaptive Servo-Ventilation (ASV) can be used to treat sleep apnea in these patients. This is an observational study to document changes in respiratory parameters in HF patients using ASV for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

More than 18 years old Chronic heart failure (at least 12 weeks since diagnosis) according to the currently applicable guidelines NYHA Class III or IV at the time of inclusion with at least one hospitalization for heart failure in the last 12 months Moderate to severe sleep apnea (AHI ≥ 15/hour). Already using or willing to use ASV-therapy and able to tolerate the mask treatment

Exclusion Criteria:

Planned or scheduled heart valve interventions and/or CABG Untreated or therapy refractory Restless Leg Syndrome Patients for whom the use of positive airway pressure therapy may be contra-indicated because of symptomatic hypotension or significant intravascular volume depletion or pneumothorax or pneumomediastinum Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Heart Failure patients using adaptive servo ventilation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Correlation of hypoxemia, as measured by overnight pulse oximetery, with worsening heart failure | 12 months
  Hypoxemia, as measured by pulse oximetery will be compared with heart failure status to measure if a correlation exists between hypoxemia and deterioration of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Oldenburg, MD, Principal Investigator — Ruhr University of Bochum
Locations (1):
- Sleep Laboratory, Ruhr University of Bochum, Bad Oeynhausen, North Rhine-Westphalia, Germany